CLINICAL TRIAL: NCT05111353
Title: Neoantigen Vaccines in Pancreatic Cancer in the Window Prior to Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Leidos (Unknown); UNICO Foundation (Unknown); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202205120
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Pancreas Cancer; Pancreatic Cancer; Cancer of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Vaccine given after neoadjuvant chemotherapy and surgery (Experimental): * The neoantigen peptide vaccine will be manufactured during neoadjuvant chemotherapy. Institutional standard of care chemotherapy will be given.
  * Peptide and poly-ICLC will be administered intramuscularly on Days 1, 4, 8, 15, 22, 50, and 78 beginning approximately 1 month after surgery. Day 1 should begin approximately 1 month after surgery.
  Interventions: Biological: Optimized neoantigen synthetic long peptide vaccine; Biological: Poly-ICLC
- Arm 2: Vaccine given after neoadjuvant chemotherapy but before surgery (Experimental): * The neoantigen peptide vaccine will be manufactured during neoadjuvant chemotherapy. Institutional standard of care chemotherapy will be given.
  * Peptide and poly-ICLC will be administered intramuscularly on Days 1, 4, 8, 15, and 22 during the chemotherapy holiday, and Days 50 and 78 post-operatively. Optimal timing for Day 1 is 1 week after end of chemotherapy, but Day 1 may be given up to 3 weeks after end of chemotherapy.
  Interventions: Biological: Optimized neoantigen synthetic long peptide vaccine; Biological: Poly-ICLC

INTERVENTIONS:
Biological: Optimized neoantigen synthetic long peptide vaccine — Neoantigen vaccines will be provided on a patient-specific basis
Biological: Poly-ICLC — Poly-ICLC will be supplied by Oncovir, Inc.
  Other Names: Hiltonol

SUMMARY:
This is a randomized phase 1 clinical trial to evaluate the safety of an optimized neoantigen synthetic long peptide (SLP) vaccines in pancreatic cancer patients following neoadjuvant chemotherapy. The neoantigen SLP vaccines will incorporate prioritized neoantigens and will be co-administered with poly-ICLC. Patients will be randomized to one of two arms: Arm 1 (neoantigen vaccine following neoadjuvant chemotherapy and surgery) or Arm 2 (neoantigen vaccine following neoadjuvant chemotherapy in the window prior to surgery).

Those who are ineligible for vaccine administration including those whose disease progresses or recurs during neoadjuvant chemo or who are otherwise unable to complete surgical resection but who had a personalized neoantigen vaccine manufactured, or significant progress has been made as determined by treating physician, are permitted to receive vaccine injections on study.

ELIGIBILITY:
Step 0 Inclusion Criteria (A patient will be eligible for evaluation and sequencing of tissue for vaccine development only if ALL of the following criteria apply:)

* Histologically or cytologically confirmed, newly diagnosed, treatment-naïve patients with localized or borderline resectable adenocarcinoma of the pancreas for whom neoadjuvant chemotherapy is considered appropriate; mixed histology (including adenosquamous). Patients with clinical suspicion of pancreatic adenocarcinoma can be enrolled for pre-treatment biopsy, and must be histologically confirmed to have adenocarcinoma before being treated on study. Patients with squamous carcinoma or neuroendocrine tumor will be excluded.
* Evaluable disease, in the opinion of the treating investigator or PI.
* Tissue specimens available in sufficient quantity to allow for sequencing.
* At least 18 years of age.
* Life expectancy of > 12 months.
* ECOG performance status ≤ 1
* Adequate bone marrow and organ function as defined below:

  * WBC ≥ 1.5 K/cumm
  * absolute neutrophil count ≥ 1.0 K/cumm
  * platelets ≥ 50 K/cumm
  * hemoglobin ≥ 8.0 g/dL
  * total bilirubin ≤ 5.0 X institutional upper limit of normal
  * AST/ALT ≤ 5.0 X institutional upper limit of normal
  * creatinine ≤2.5 X institutional upper limit of normal OR creatinine clearance ≥ 30 mL/min by Cockcroft-Gault for patients with creatinine levels above institutional normal
  * Note: labs can be repeated prior to chemo if needed.
  * Note: Patients who have had a stent placed for biliary obstruction and whose liver function is expected to improve may enroll provided serum bilirubin at time of enrollment is within the limits above.
* International Normalized Ratio (INR) and activated partial thromboplastin time (PTT) < 2.0 x ULN provided the patient is not on anticoagulation therapy.
* Women of childbearing potential and men must agree to use two forms of adequate contraception prior to study entry, for the duration of study participation, and for 3 months after completion of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document.

Step 0 Exclusion Criteria (A patient will be eligible for evaluation and sequencing of tissue for vaccine development only if ALL of the following criteria apply:)

* Evidence of predominantly neuroendocrine (defined by > 50% histology) tumor, pure neuroendocrine tumor, duodenal adenocarcinoma, or ampullary adenocarcinoma.
* History of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only, carcinoma in situ of the cervix, or LCIS/DCIS of the breast.
* Receiving any other investigational agents, or planning to receive other investigational agents as part of neoadjuvant therapy.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, hepatic renal, and/or other functional abnormality that might jeopardize the health and safety of the participant as determined by the investigator based on medical history, physical examination, laboratory values, and/or diagnostic studies. If needed and appropriate. the final determination related to study eligibility prior to the administration of the first vaccine will be documented by both the PI and Sub-Investigators in consultation with a specialist.
* A psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator from the medical history, physical exam, and/or medical record
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. In the case of asthma or chronic obstructive pulmonary disease taking inhaled corticosteroids that does not require daily systemic corticosteroids is acceptable. Additionally, local acting steroids (topical, inhaled, or intraarticular) will be allowed. Patients on intermittent or short course steroids will be allow if the dose does not exceed 4 mg of dexamethasone (or equivalent) per day for > 7 consecutive days. Premedication for chemotherapy does not apply to this criteria and may be administered as per SOC practice. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant and/or breastfeeding.
* Known HIV-positive status.
* History of positive test for Hepatitis B virus surface antigen (HBsAg) and/or positive Hepatitis C antibody result with detectable hepatitis C virus (HCV) ribonucleic acid (RNA) indicating acute or chronic infection.

Step 1 Eligibility: At Step 1 eligibility confirmation prior to vaccination, the above criteria must be met plus:

* Completed at least 4 months of neoadjuvant chemotherapy such as FOLFIRINOX, modified FOLFIRINOX, or gemcitabine + nab-paclitaxel. Dose modifications and/or delays in neoadjuvant chemotherapy may be made at the discretion of the treating physician
* Reimaging within 4 weeks of last dose of chemotherapy demonstrates no evidence of progressive disease. Patients who progress on mFOLFIRINOX and transition to gemcitabine + nab-paclitaxel may still be eligible for vaccine administration at discretion of PI and treating MD provided they do not show progression following completion of chemotherapy and the patient continues to be eligible for surgical resection. Patients who, in the opinion of the treating physician, require SBRT prior to surgery will receive vaccine after surgery regardless of randomization.

  **Patients who progress or recur following neoadjuvant chemotherapy or who are otherwise unable to complete a surgical resection, but who still meet other Step 1 criteria, may still be eligible for vaccine administration with documented treating physician and PI approval.
* There is a 1 week washout prior to Day 1 of vaccine for patients on daily systemic steroids at doses exceeding 10 mg prednisone.
* Must not be receiving or have received any other investigational agents within the last 30 days. Note that patients who are receiving or will be receiving adjuvant chemotherapy are permitted to continue on study and are considered eligible.
* Patients may not have received a live vaccine within 30 days prior to the first day of treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Sufficient wound healing per the evaluation of the treating physician.
* If a patient experiences disease progression or recurrence during neoadjuvant chemotherapy, or is otherwise unable to complete a surgical resection after sufficient progress has been made on the vaccine production, the participant may still receive treatment with the peptide vaccine. Eligibility for continued participation in these cases will be at the treating physician and PI's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Safety of neoantigen SLP vaccine as measured by number of subjects experiencing each type of adverse event | Through 4 weeks after completion of last vaccination (estimated to be 108 days)
  -Adverse events will be characterized according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (CTCAE).

SECONDARY OUTCOMES:
Immunogenicity of neoantigen peptide vaccine as measured by the the number of neoantigen-specific T cells (only Arm 1 and Arm 2) | Through approximately 2 years and 78 days
  * Immune monitoring will occur at baseline, at time of surgery, day 1, day 15, day 22, day 50, and day 78 for Arm 1. Optional monitoring at 1 and 2 years after last vaccine administration
  * Immune monitoring will occur at baseline, day 1, day 15, day 22, day 50, at the time of surgery, and day 78 for Arm 2. Optional monitoring at 1 and 2 years after last vaccine administration.
Immunogenicity of neoantigen peptide vaccine as measured by the phenotype of neoantigen-specific T cells (only Arm 1 and Arm 2) | Through approximately 2 years and 78 days
  * Immune monitoring will occur at baseline, at time of surgery, day 1, day 15, day 22, day 50, and day 78 for Arm 1. Optional monitoring at 1 and 2 years after last vaccine administration
  * Immune monitoring will occur at baseline, day 1, day 15, day 22, day 50, at the time of surgery, and day 78 for Arm 2. Optional monitoring at 1 and 2 years after last vaccine administration.

CONTACTS AND LOCATIONS:
Overall Officials: William E Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data will be submitted to the database of Genotypes and Phenotypes (dbGap) at the National Cancer Institute.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu